CLINICAL TRIAL: NCT04352855
Title: Ceftolozane-tazobactam for the Treatment of Respiratory Infections Due to Extensively Drug-resistant Pseudomonas Aeruginosa Among Critically Ill Patients: a Retrospective Study.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Zsolt Iványi, Associate professor, Semmelweis University
Other Study IDs: SE58/2020
Record Dates: First submitted 2020-04-15; First posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Ventilator Associated Pneumonia; Antibiotic Resistant Infection
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — ceftolozane, tazobactam drug combination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- C/T: C/T cases: individuals fulfilling eligibility criteria and treated with ceftolozane-tazobactam
  Interventions: Drug: Ceftolozane/tazobactam
- C: C cases: individuals fulfilling eligibility criteria and treated with colomycine

INTERVENTIONS:
Drug: Ceftolozane/tazobactam — Administration
  Groups: C/T

SUMMARY:
The aim of this study is to report our experience with ceftolozane-tazobactam and to evaluate its safety and efficacy in the treatment of ICU dependent nosocomial respiratory tract infections due to extensively drug resistant Pseudomonas aeruginosa. Different dosing regimes of ceftalozane-tazobactam is evaluated and compared to the standard therapy of Colomycin.

DETAILED DESCRIPTION:
Ceftolozane-tazobactam (C/T) is a novel type of beta-lactam/beta-lactamase inhibitor antibiotics targeting nosocomial infections caused by Gram-negative bacteria. In recent years, ceftolozane-tazobactam was prescribed for treating complicated urinary tract infections (cUTI) and complicated intraabdominal infections (cIAI). Following the results of ASPECT-NP trial in 2019, it was approved as a therapeutic option in nosocomial pneumonia including hospital-acquired pneumonia (HAP) and ventilator-associated pneumonia (VAP).

The drug shows an excellent activity against ESBL-producing Enterobacterales and multidrug-resistant (MDR) and extensively drug-resistant (XDR) strains of Pseudomonas aeruginosa. The latter is widely recognized as a common pathogen of nosocomial respiratory tract infections.

There is still a need for observations of clinical experiences to better define the risk-benefit profile of ceftolozane-tazobactam. The aim of this study is to report our experience with ceftolozane-tazobactam and to evaluate its safety and efficacy in the treatment of ICU dependent nosocomial respiratory tract infections due to extensively drug resistant Pseudomonas aeruginosa. Different dosing regimes of ceftalozane-tazobactam is evaluated and compared to the standard therapy of Colomycin.

ELIGIBILITY:
Inclusion Criteria:

* Hospital-acquired pneumonia caused by extensively drug-resistant Pseudomonas aeruginosa
* ≥ 72 hours of targeted antibiotic therapy against Pseudomonas aeruginosa with either Colomycin or Ceftolozane-Tazobactam

Exclusion Criteria:

* Participation in an interventional trial aiming nosocomial infections
* Treatment was not with the intent to cure the infection

Ages: 16 Years to 90 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to a multideisciplanry academic terciary care ICU, suffering from ventilation associated pneumonia, caused by XDR or panresistant Pseudomonas Aeruginosa
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2020-05-19 (Estimated); Study Completion 2020-05-19 (Estimated)

PRIMARY OUTCOMES:
Clinical cure rate | 7-14 day
Microbiological cure rate | 7-14 day

SECONDARY OUTCOMES:
LOS | 28
  Lenght of ICU stay
Length of ventilation | Untill patient is ventilated (expected time frame is 10 days)
28 day mortality | 28
Drug related adverse events rate | until ICU discharge (expected average day is 14)
  The number and nature

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No